CLINICAL TRIAL: NCT03471091
Title: Effect of the Integrated Network Management of Stable Hypercapnic COPD Patients With Domiciliary Noninvasive Ventilation Treatment
Brief Title: Clinical Evaluation of COPD Butler in Patient Home Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Guangdong Second Provincial General Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Guangzhou First People's Hospital (Other); Dongguan People's Hospital (Other Government); Huizhou Municipal Central Hospital (Other); Shenzhen People's Hospital (Other); Clifford Hospital, Guangzhou, China (Other); Shenzhen Sixth People's Hospital (Other); Subei People's Hospital of Jiangsu Province (Other)
Responsible Party: Principal Investigator, Rongchang Chen, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GIRH-201801
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: COPD; Hypercapnic Respiratory Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group subjects will use NIV with the integrated tele-monitoring management program as home therapy and accomplish the following tasks via mobile COPD Butler APP: 1) upload daily NIV usage data， blood pressure, oxygen saturation, and heart rate measurement; 2) daily medication taken recording; 3) regular self-reported health questionnaire and symptom recording; 4) read health education materials.
  Information collected from the intervention group by the APP will be monitored by physician team from the leading hospital through physician web portal. The physician team will provide regular health report, and once an alert is generated due to the abnormality in NIV usage or vital sign data etc., physicians will take action accordingly.
  Interventions: Device: NIV with the integrated tele-monitoring management program
- Control group (No Intervention): Control group subjects will only use NIV according to their treatment plan at home. NIV usage data will be read from the NIV secure digital memory card for the control group.

INTERVENTIONS:
Device: NIV with the integrated tele-monitoring management program — Noninvasive positive pressure ventilation with the integrated tele-monitoring management will provide regular health report, and once an alert is generated due to the abnormality in NIV usage or vital sign data etc., physicians will take action accordingly.
  Arms: Intervention group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a worldwide common disease with high morbidity and mortality and leads to heavy social and economic burden. Health management of stable COPD patients has been suggested to be essential for delaying diseases progress, reducing acute exacerbation events and improving patient quality of life. Non-invasive ventilation (NIV) is a widely used treatment in COPD patients. There were studies shown that NIV could improve ventilation, blood gases etc., and several clinical trials have shown improvements in survival, exercise capacity, quality of life and so on. Compliance to NIV and optimal parameter setting are important factors that will affect the effect of the use of NIV, thus NIV usage monitoring might also be a crucial element in the health management of COPD patients. Many studies have been designed to study the effect of tele-monitoring program on the management of COPD patients. However, almost none of these studies were designed for specific population, and little is known about the effect of such program on the management of patients with NIV treatment.

DETAILED DESCRIPTION:
The COPD home management program consists of 3 Philips devices (NIV BiPAP ST, Oximeter and Blood Pressure Meter), a patient mobile APP which is developed for self-management at home and a professional physician web portal which is designed for NIV usage and other vital sign data monitoring. The program is intended to manage the post-discharge COPD patient by enhancing COPD patient condition monitoring and adherence to the home therapy, e.g. NIV in this study. Besides obtaining clinical proof points of the efficacy of such program on patients with NIV treatment, it will provide potential evidence of the usability as well as the collect the insights for future product improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80, males and females
2. Stage III and IV COPD
3. Daytime hypercapnia (PaCO2 ≥ 50 mmHg) at rest without ventilatory support
4. Possess home oxygen concentrator
5. Participants/Caregivers have access to and capable of using smartphone and internet
6. Willing to participate in the study
7. Able to provide informed consent

Exclusion Criteria:

1. Subjects with NIV as routine therapy prior to the study
2. Subjects with abnormalities of the lung or thorax other than COPD
3. Subjects with obstructive sleep apnea, COPD with obstructive sleep apnea overlap syndrome, severe heart failure, severe arrhythmias, unstable angina, and malignant comorbidities
4. Subjects with significantly impaired cognitive function and are unable to fulfill the study requirement (unable to provide informed consent)
5. Subjects who participated in another trial within 30 days prior to the planned start of study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to NIV treatment | 12th month
  The primary objective is to test the effect of COPD tele-monitoring program on patient's adherence to NIV treatment.

SECONDARY OUTCOMES:
Acute exacerbation of COPD re-admission rate | Baseline, 1st, 3rd, 6th and 12th month
  Acute exacerbation which was characterized as an acute worsening of more than one respiratory symptom (new onset of or increase in sputum volume or purulence, wheezing, cough, dyspnoea, or fever) lasting for at least 2 consecutive days and result in any changes in their conventional therapy.
Severe Respiratory Insufficiency (SRI) Questionnaire | Baseline, 3rd, 6th and 12th month
  The SRI Questionnaire has good psychometric properties shown to be valid for chronic hypercapnic COPD patients receiving NIV. It includes 49 items on seven subscales.
COPD assessment test | Baseline, 1st, 3rd, 6th and 12th month
  The COPD Assessment Test is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time.
Partial pressure of arterial blood carbon dioxide (PaCO2) | Baseline, 1st, 3rd, 6th and 12th month
  Daytime arterial blood gas samples were taken with patients resting in a sitting position and breathing room air without having used NIV for at least 1 hour.
6-minute walk test | Baseline, 3rd, 6th and 12th month
  The 6-minute walk test plays a key role in evaluating functional exercise capacity, assessing prognosis and evaluating response to treatment across a wide range of respiratory diseases.
Forced vital capacity | Baseline, 3rd, 6th and 12th month
  Forced vital capacity is measured in a test known as spirometry, a type of pulmonary function test, which is used to help determine both the presence and severity of lung diseases.
Forced expiratory volume in 1 second | Baseline, 3rd, 6th and 12th month
  Forced expiratory volume in 1 second is a marker used to measure lung function and can help you monitor your lung diseases over time.
Baseline Dyspnea Index/Transition Dyspnea Index | Baseline, 3rd, 6th and 12th month
  Baseline Dyspnea Index/Transition Dyspnea Index provides a multidimensional measurement of dyspnea based on 3 components that evoke dyspnea in activities of daily living, in symptomatic individuals.
COPD self-efficacy scale | Baseline, 6th and 12th month
  Identifying situations in which individuals with COPD experience low self-efficacy is important.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, MD, Study Director — Guangzhou Institute of Respiratory Health
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University., Guangzhou, Guangdong, China